CLINICAL TRIAL: NCT05207449
Title: Health Challenges for Adolescents With Chronic Diseases Attending Assiut University Children Hospital and Sidi Galal Health Insurance Clinic
Brief Title: Health Challenges for Adolescents With Chronic Diseases in Egypt
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam Gamal, Principle investigator, Assiut University
Other Study IDs: PhD2021
Record Dates: First submitted 2021-09-06; First posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Adolescent Behavior; Chronic Disease; Adherence, Medication; Quality of Life
MeSH Terms: conditions — Adolescent Behavior; Chronic Disease; Medication Adherence | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — The questionnaire will include:
  1. The demographic data of the patients
  2. Chronic disease related questions
  3. Assessment of adherence to treatment by using Arabic validated version of Medication Adherence Report Scale (MARS)
  4. Patients' beliefs about medication will be assessed using Arabic validated version of Beliefs about Medicines Questionnaire (BMQ)
  5. Disease acceptance will be evaluated using: Arabic validated version of Acceptance to Illness Scale (AIS)
  6. Assessment of health-related quality of life (HRQoL) using the Arabic version of the Pediatric Qualify of Life Inventory Generic Core Scale (PedsQL) 4.0 GCS
  7. Assessment of readiness for transition to adult health care settings using The Transition Readiness Assessment Questionnaire (TRAQ)

SUMMARY:
The World Health Organization (WHO) defines adolescents as those people between 10 and 19 years of age. Adolescence is a critical developmental stage especially in the context of living with a chronic disease (CD), a chronic disease can be defined as "physiological, behavioral or cognitive disorder that has lasted for one year and produces one or more types of consequences: functional constraints, dependency on compensatory assistance for functioning, or increased need of service compared with age-mates".

The burden of chronic conditions in adolescence is increasing as larger numbers of chronically ill children survive beyond the age of 10. Over 85% of children with congenital or chronic conditions now survive into adolescence, and conditions once seen only in young children are now seen beyond childhood and adolescence.

DETAILED DESCRIPTION:
Adolescents live a complex period of their lives, where several unique transformations take place (urge for personal identity, autonomy and independence), having a chronic condition in this period can represent an additional burden for those natural developmental challenges.

In fact, The developmental processes involved in adolescence have a complex and bi-directional interaction with chronic illness such that a chronic disease can alter development and vice versa. For example, some chronic diseases, such as cystic fibrosis or diabetes mellitus, can impair pubertal development. On the other hand, puberty itself can affect the course of a chronic disease. For example, normal puberty is associated with insulin resistance; therefore, blood glucose control can be difficult during pubertal years in teens with diabetes.

Unlike adults, adolescents with chronic disease find more difficulties facing challenges as adherence to treatment, impaired quality of life, disease acceptance and eventually transition to adult health care settings.

Adherence to treatment:

Adherence to treatment is defined as "the extent to which a person's behavior, in terms of taking medications, following diets, or executing lifestyle changes, coincides with medical or health advice".

Low adherence to treatment is common in adolescents and it increases morbidity and medical complications, contributes to poorer quality of life and an overuse of the health care system, particularly during the transition from pediatric health care to adult-centered health care.

There are many factors affecting adherence to treatment in adolescents such as demographic, familial, socioeconomic, personal, type of illness, therapeutic regimens and the relationship with health care professionals. Also, patient's beliefs, concerns and attitudes toward medication are considered among the most important drivers of non-adherence among chronic disease patients as several studies have shown that patients who have concerns and negative attitudes towards their medications are less adherent than those who have positive beliefs and attitude .

Health related quality of life (HRQoL):

Survival from chronic diseases in adolescence has globally increased in the last decades, due to advances in pediatric medicine and in life expectancy at birth. However, surviving is not sufficient but rather the quality of survival, so health-related quality of life (HRQOL) issues have become more important.

Adolescents may feel that living with a chronic health condition impair physical, cognitive, social and emotional dimensions, as well as general quality of life (QoL) and health-related quality of life (HRQoL).

HRQoL is a more restricted concept that focuses on the impact of health and illness on the individual's QoL and overall well-being. The concept of HRQoL was introduced in healthcare as a specific component of the broader QoL construct, comprehending the subjective impact of health conditions, medical treatments and healthcare policies. It is considered closer to the concept of "disease impact" and theoretically distinct from the QoL wider construct (although it is still related).

The last decade has evidenced a dramatic increase in the development and utilization of pediatric HRQOL measures in an effort to improve patient health and well-being and to determine the value of healthcare services. A generic HRQOL instrument must be multidimensional, consisting at the minimum of the physical, psychological (including emotional and cognitive), and social health dimensions delineated by the World Health Organization.

Acceptance of disease:

In the context of chronic illness, it has been suggested that the way in which adolescents accept their illness plays an important role in their well-being. Acceptance can be defined as 'recognizing the need to adapt to chronic illness while perceiving the ability to tolerate the unpredictable, uncontrollable nature of the disease and handle its averse consequences'. In other words, Acceptance is conceptualized as the perceived ability to live with the illness and to master its negative consequences. Higher acceptance of chronic illness is related to positive outcomes such as less anxiety, less depression, less disability and better emotional, social and physical functioning.

Research has shown that young people who could focus on the positive aspects of their condition had more favorable treatment outcomes and recovery from illness compared to those who did not.

Transition to adult health care:

As a large number of children with chronic conditions now reach adulthood; accompanied by significant ongoing healthcare needs related to their chronic condition, so the issue of the transition from the paediatric setting to the adult setting has become a fundamental focus of comprehensive healthcare. consequently, the process and organization of transition is becoming increasingly important.

Transition is defined as the purposeful, planned movement from paediatric to adult medicine upon entering adulthood. The multidimensional nature of the transition process includes medical as well as psychosocial and educational/vocational issues.

There is increasing evidence that an unsuccessful transition due to missing follow-up care through a clinical specialist in adult medicine may result in discontinuity in treatment, a decrease in doctors' visits or an increase in changing physicians and in poor health outcomes.

The optimal age of transition is still debated and thus requires further investigation in transition research. In a systematic review of the research on transition, the optimal age range of transfer in 14 of the 15 papers was 18-19 years. However, some other studies have shown that the timing of transition should be based on the level of maturity and responsibility, and not on chronological age. The American Academy of Pediatrics (AAP) advises that parents and their doctors begin to plan for transition as early as age 12.

Patient education programmes and skills training that enhance self-management and empowerment can prepare adolescents for this complex transition process. It is emphasized that 'strengthening adolescents' independence and self-management competencies, combined with early preparation and repeated discussions about the forth- coming transition, seem to be a useful strategy in increasing adolescents' readiness to transfer'. It's argued that a generic patient education programme may be useful because psychosocial issues associated with the transition process are similar and often independent of the diagnosis .

ELIGIBILITY:
Inclusion Criteria:

* Any adolescent aged 10-18 years having chronic disease for more than one year with regular medications prescriptions

Exclusion Criteria:

-

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents with different chronic disease (such as: DM-1, thalassemia, rheumatoid arthritis, systemic lupus and chronic kidney disease, etc..) attending different pediatric outpatient clinics and inpatient units at Assiut University Pediatric Hospital and Sidi Galal Health Insurance Clinic.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of adolescents with chronic conditions showing good adherence to treatment as measured by Medication Adherence Report Scale (MARS) | 6 months
  3- Assessment of adherence to treatment by using Arabic validated version of Medication Adherence Report Scale (MARS): 5- items rated on a 5-point scale.
  The cut point used for the MARS score will be ≥80% (i.e. if the score ¬≥ 20 the adolescent will be considered adherent)
percentage of adolescents with chronic disease showing high acceptance to thier chronic disease measured by Acceptance to Illness Scale (AIS) | 6 months
  5- Disease acceptance will be evaluated using:
  Arabic validated version of Acceptance to Illness Scale (AIS) (42) which consists of 8- items rated on a 5-point scale, where (1 means strongly agree; 2-agree; 3-undecided; 4-disagree; 5-strongly disagree) .
  The total score of the scale ranges from 8 to 40; the higher score, the better acceptance of illness.
percentage of adolescents with chronic disease showing high quality of life measured by Arabic version of the Pediatric Qualify of Life Inventory Generic Core Scale | 6 months
  6- Assessment of health-related quality of life (HRQoL) using the Arabic version of the Pediatric Qualify of Life Inventory Generic Core Scale (PedsQL) 4.0 GCS (43):
  It is a 23-item which includes:
  1. Physical Functioning (8 items).
  2. Emotional Functioning (5 items).
  3. Social Functioning (5 items).
  4. School Functioning (5 items).
  The response options of the PedsQL (4.0) require children to rate each item using a 5-point rating scale ranging from 'never' to 'almost always' as follow:
  * 0 if it is never a problem.
  * 1 if it is almost never a problem.
  * 2 if it is sometimes a problem.
  * 3 if it is often a problem.
  * 4 if it is almost always a problem Each item was then reverse scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, 4=0, so that higher scores indicate a better HRQoL
Percentage of adolescents with chronic disease showing high readiness for transition to adult health care setting measured by The Transition Readiness Assessment Questionnaire (TRAQ) | 6 months
  7- Assessment of readiness for transition to adult health care settings using The Transition Readiness Assessment Questionnaire (TRAQ), which is a validated 20-item, 5-domain (appointment keeping- tracking health issues- managing medications-taking with providers-managing daily activities) patient-reported assessment of health and health care self-management skills that can be used in preparation for transition to adult care

IPD SHARING:
Plan to Share IPD: Undecided